CLINICAL TRIAL: NCT06419244
Title: Myosteatosis in Oeso-gastric Cancer: Clinical Impacts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: TuMECA
Record Dates: First submitted 2024-03-20; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Cancer; Gastric Cancer; Myopenia; Adipose Tissue Tumor
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Neoplasms, Adipose Tissue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical patients (Other): Patients undergoing surgery
  Interventions: Diagnostic Test: Myosteatosis
- Non surgical patients (Other): Patients not undergoing surgery
  Interventions: Diagnostic Test: Myosteatosis

INTERVENTIONS:
Diagnostic Test: Myosteatosis — Determination of myosteatosis by imaging

SUMMARY:
The aim of this project is to study the presence of cancer-associated adipocytes in oesogastric cancers and their possible links with myosteatosis. This research project has a retrospective component, the aim of which is to analyse the body component based on imaging in patients with oesogastric neoplasia in order to determine the incidence of myosteatosis and to study the relationship with oncological and prognostic data. The second part of the project is prospective and will collect biological material (skeletal muscle, adipose tissue, tumour, blood) for histological, molecular and genomic analyses and will analyse muscle function in patients with oesogastric cancer. It will address the role of adipocytes in the tumour microenvironment of oesogastric cancer, focusing on their interactions with the observed muscle myosteatosis and prognosis. In the future, it will help to identify signalling pathways, targets and patients who could benefit from appropriate treatment.

DETAILED DESCRIPTION:
Oesophageal and gastric cancer pose a significant challenge to caregivers, both in terms of the complexity of its presentation and its treatment. At diagnosis, patients often present with malnutrition associated with sarcopenia, which has a significant impact on morbidity and mortality. Although loss of muscle mass has received much attention in cancer, muscle quality, particularly the accumulation of fat in muscle named "myosteatosis", may be considered as a better predictor of a patient's physical condition and ability to recover from cancer treatments. Studying the tumor microenvironment is essential to understanding the mechanisms underlying disease progression. Cancer-associated adipocytes (CAA), a major component of this tumor microenvironment, provide an interface for dialogue with the tumor through the secretion of pro-inflammatory cytokines, metalloproteases and the release of free fatty acids. They have been described as capable of stimulating tumor progression, particularly in breast cancer. However, their presence in oesogastric cancer and possible links with myosteatosis have not been described.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer of the oesophagus, oeso-gastric junction or stomach
* Treatment and estimated survival of more than 3 months
* Signed informed consent
* > 18 years of age

Exclusion Criteria:

* Neuromuscular or orthopedic pathology
* Cognitive disorders
* Psychiatric disorders
* Inability to communicate in French or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Myosteatosis | Through study completion, an average of 2 years
  Muscle fat infiltration measured by analysis of tissue density based on a CT scan in L3 with the help of body component analysis software

SECONDARY OUTCOMES:
Physical functional status 1 | Through study completion, an average of 2 years
  Hand grip test
Physical functional status 2 | Through study completion, an average of 2 years
  6 minutes walking test
Physical functional status 3 | Through study completion, an average of 2 years
  Chair lift test
Cancer-associated adipocytes | Through study completion, an average of 2 years
  Determining the presence and impact of tumor-associated adipocytes

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Deswysen, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No